CLINICAL TRIAL: NCT07160634
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy of a Single Intravenous Dose of SGT-003 in Ambulant Males With Duchenne Muscular Dystrophy
Brief Title: A Study of SGT-003 Gene Therapy in Ambulant Males With Duchenne Muscular Dystrophy (IMPACT DUCHENNE)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Solid Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGT-003-301; 2025-522949-22 (EudraCT Number); 1013075 (Other: IRAS)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: SGT-003; Duchenne Muscular Dystrophy (DMD); adeno-associated virus (AAV); IMPACT DUCHENNE
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SGT-003 followed by Placebo (Experimental): Enrolled participants will receive a single intravenous (IV) infusion of SGT-003 in Part 1 and a single IV infusion of matching Placebo in Part 2.
  Interventions: Drug: SGT-003; Drug: Placebo
- Placebo followed by SGT-003 (Experimental): Enrolled participants will receive a single intravenous (IV) infusion of matching Placebo in Part 1 and a single IV infusion of SGT-003 in Part 2.
  Interventions: Drug: SGT-003; Drug: Placebo

INTERVENTIONS:
Drug: SGT-003 — Adeno-associated virus (AAV)-based gene therapy that delivers a codon-optimized and CpG island-minimized human 5-repeat microdystrophin (h-μD5)
Drug: Placebo — IV infusion

SUMMARY:
This is a Phase 3, double-blind, placebo-controlled study with the primary objective of evaluating the efficacy of a single IV infusion of SGT-003 in pediatric ambulant male participants with DMD. The secondary objectives include the evaluation of additional efficacy and safety outcomes. The study will be divided into 2 parts. Participants will be randomized 1:1 to either SGT-003 in Part 1 followed by placebo in Part 2 or to placebo in Part 1 followed by SGT-003 in Part 2. Participants will continue to be monitored in long term follow up (LTFU) for at least 5 years from their SGT-003 dosing date.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ambulatory.
* Established clinical diagnosis of DMD and documented DMD gene mutation predictive of DMD phenotype.
* Negative for antibodies against adeno-associated virus.
* On a stable daily oral regimen of at least 0.5 mg/kg/day prednisone or 0.75 milligrams per kilogram per day (mg/kg/day) deflazacort for at least 6 months prior to entering the study, allowing for weight-based dose modifications in accordance with clinical practice.
* Meet 10-meter walk/run time criteria.
* Meet time to rise from supine criteria.
* Participant has bodyweight ≤50 kg.

Exclusion Criteria:

* Current or prior treatment with an approved or investigational gene transfer drug or gene editing therapy.
* Exposure to vamorolone, givinostat, approved or investigational dystrophin- or disease-modifying drugs (such as eteplirsen, golodirsen, casimersen, viltolarsen, and ataluren), or another investigational drug for any indication within 6 months or 5 half-lives, whichever is longer, prior to enrollment.
* Established clinical diagnosis of DMD that is associated with any deletion variant or variant predicted not to express exons 1 to 11, exons 42 to 45, or exons 57 to 69, inclusive of the DMD gene as documented by a genetic report.

Other Inclusion/Exclusion criteria to be applied as per protocol.

Ages: 7 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Time to Rise (TTR) from Supine Velocity (rise/s) at Day 540 | Baseline, Day 540

SECONDARY OUTCOMES:
Change From Baseline in Stride Velocity 95th Centile (SV95C) (m/s) at Day 540 | Baseline, Day 540
Change From Baseline in 4-Stair Climb (4SC) Velocity (tasks/s) at Day 540 | Baseline, Day 540
Change From Baseline in 10-meter Walk/Run (10MWR) Velocity (m/s) at Day 540 | Baseline, Day 540
Change From Baseline in North Star Ambulatory Assessment (NSAA) total score at Day 540 | Baseline, Day 540
Cumulative Loss of Function in NSAA Items at Day 540 | At Day 540
Change From Baseline in Microdystrophin Protein Levels by western blot (% of normal dystrophin) at Day 90 | Baseline, Day 90
Change From Baseline in Microdystrophin Tissue Distribution by Immunofluorescence (% positive fibers) at Day 90 | Baseline, Day 90
Change from baseline in Percent Predicted Forced Vital Capacity (FVC) at Day 540 | Baseline, Day 540
Change from baseline in Percent Predicted Peak Expiratory Flow (PEF) at Day 540 | Baseline, Day 540
Change from baseline in Percent Predicted Forced Expiratory Volume in 1 second (FEV1) at Day 540 | Baseline, Day 540
Change from baseline in the Pediatric Outcomes Data Collection Instrument (PODCI) Global score at Day 540 | Baseline, Day 540
Number of Participants with Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Adverse Events of special interest (AESIs), and clinically significant changes in Electrocardiogram (ECG) and Echocardiography (ECHO) | From first dose up to Day 540

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No